CLINICAL TRIAL: NCT06187246
Title: An Avatar-based Intervention in Second Life for Female Orgasmic Disorder: A Randomized Control Trial
Brief Title: Avatar-based Therapy for Female Orgasmic Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Ariana Vila, Principal investigator, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UniversidadRJC 2005202114121
Record Dates: First submitted 2023-12-05; First posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Female Orgasmic Disorder

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Avatar-based Intervention Group (Experimental): Treatment was based on the CBT approach and previous literature about FOD. It consisted of 12 weekly online individual sessions, which were administered once a week (total duration = 3 months) and lasted about 60 minutes each.
  Interventions: Behavioral: Avatar-based intervention
- Minimal support control group (Active Comparator): It consisted in individual informative talks, during which they were provided with information about female orgasm (e.g., what is an orgasm, neuronal orgasm, factors that may influence consecution, sexual response), masturbatory techniques (e.g., key elements to achieve pleasure, anatomy of the female genitalia, pleasure areas) and techniques to focus attention on one's body (i.e., an important factor to pleasure). Participants received three individual sessions once a month, and had a duration of one hour.
  Interventions: Other: Individual informative talks

INTERVENTIONS:
Behavioral: Avatar-based intervention — Intervention was aimed at improving sexual variables (sexual satisfaction, sexual function, and initiative and sexual communication), and variables that are known to affect orgasm consecution (sexual self-esteem, sex-guilt, and sexual anxiety). To achieve this objective, it focused on fostering participants' abilities to increase their levels of sexual stimulation, and the engagement in personal values, along with identifying and modifying dysfunctional thoughts about sexuality. The techniques used included psychosexual education, cognitive restructuring, virtual exposure, sexual stimulation, and engagement in personal values from the acceptance and commitment therapy (ACT) perspective.
  It was delivered via a metaverse: Second Life.
  Arms: Avatar-based Intervention Group
Other: Individual informative talks — Participants were provided with information about female orgasm (e.g., what is an orgasm, neuronal orgasm, factors that may influence consecution, sexual response), masturbatory techniques (e.g., key elements to achieve pleasure, anatomy of the female genitalia, pleasure areas) and techniques to focus attention on one's body (i.e., an important factor to pleasure). Participants received three individual sessions once a month, and had a duration of one hour.
  Arms: Minimal support control group

SUMMARY:
A randomized controlled trial was conducted for testing the efficacy of a novel avatar-based intervention (IG), that was compared with a control group (CG) for women with female orgasmic disorder (FOD). Participants were 31 women who were randomly assigned to the intervention or the control conditions. Intervention was based on the cognitive behavioral therapy approach (treatment with the most empirical evidence) and previous literature about FOD. It consisted of 12 weekly online individual sessions and aimed at improving the FOD diagnosis, sexual variables, and variables that are known to affect orgasm consecution. Control group was based on minimum therapeutic contact. Changes over time in the assessed variables were analyzed using linear mixed models, considering treatment group, measurement time point, and group-by-time interactions as fixed effects. Effect sizes were computed (Cohen's d; number needed to treat - NNT; reliable change index - RCI).

ELIGIBILITY:
Inclusion Criteria:

* Present the characteristics to diagnose female orgasm disorder after a clinic assessment (considering natural characteristics of the women's sexual response cycle (Conn & Hodges, 2022) based on the DSM-5 criteria.
* Provide a medical check to prove the absence of physical factors that may be the cause of the orgasm dysfunction, as this is the first part to diagnose FOD.
* Be at least 18 years old (adult).
* Have access to a computer with the characteristics to run Second Life and internet connection.

Exclusion Criteria:

* Present a diagnosis of a physical condition that may be the cause of the orgasm dysfunction (e.g., genital lesions, systemic and hormonal factors, vulvovaginal atrophy).
* Presence of other psychological pathology (e.g., depression, trauma) that may be the cause of the orgasm dysfunction.
* Have alcohol dependence (i.e., evaluated during the clinical assessment, according to the diagnostic criteria from the DSM-5, to determine if the individual meets the criteria for an alcohol use disorder diagnosis).
* Drug use, including medication that is known to cause sexual difficulties (e.g., selective serotonin reuptake inhibitors (SSRIs), that are a particularly common drug cause of sexual dysfunction.
* Have participated in a previous psychological intervention in the last year.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Sexual satisfaction assessed by the Golombok Rust Inventory of Sexual Satisfaction | From baseline to the end of the treatment at 12 weeks + 1 month-follow-up and 3 month-follow-up
  Sexual satisfaction is the feeling of pleasure that one has when the sexual desire has been fulfilled.
  The Golombok Rust Inventory of Sexual Satisfaction has minimum-maximum values of 0-112; higher scores mean a worse outcome. The cut-off for determining significant levels of Sexual Satisfaction is 60 (scores equal to or above 60 indicate the existence of a sexual problem).
Sexual functionassessed by the Female Sexual Function Index | From baseline to the end of the treatment at 12 weeks + 1 month-follow-up and 3 month-follow-up
  Sexual function refers to the capacity of having a satisfactory sexual life. The Female Sexual Function Index has minimum-maximum values of 19-95; higher scores mean a better outcome. The cut-off for determining signiﬁcant levels of this variable is 55 (scores equal to or below 55 indicate poor Sexual Function).
Initiative and Sexual Communication assessed by the Female Sexual Function Questionnaire | From baseline to the end of the treatment at 12 weeks + 1 month-follow-up and 3 month-follow-up
  Initiative and Sexual Communication is the proactive and consensual expression of one's sexual desires, interests, and intentions within the context of a sexual relationship or encounter.
  The Female Sexual Function Questionnaire has minimum-maximum values of 14-70; higher scores mean a better outcome. The cut-off for determining significantly low levels of this variable are scores equal to or lower than 25.

SECONDARY OUTCOMES:
Sexual self-esteem assessed by the Rosenberg Self-Esteem Scale | From baseline to the end of the treatment at 12 weeks + 1 month-follow-up and 3 month-follow-up
  Self-esteem related to sexuality; may influence on the consecution of orgasms. The Rosenberg Self-Esteem Scale has minimum-maximum values of 10-40; higher scores mean a better outcome. The cut-off for clinical low self-esteem is a score equal to or lower than 25.
Sex-guilt assessed by the Brief Mosher Sex-Guilt Scale | From baseline to the end of the treatment at 12 weeks + 1 month-follow-up and 3 month-follow-up
  Sex-guilt related to sexuality; may influence on the consecution of orgasms. The Brief Mosher Sex-Guilt Scale has minimum-maximum values of 10-60; higher scores mean a worse outcome (higher scores indicate higher levels of guilt).
Sexual anxiety by the Sexual Anxiety scale of the Expanded Sexual Arousability Inventory | From baseline to the end of the treatment at 12 weeks + 1 month-follow-up and 3 month-follow-up
  Sexual anxiety related to sexualiaty; may influence on the consecution of orgasms.
  TheSexual Anxiety scale of the Expanded Sexual Arousability Inventory has minimum-maximum values of 0-168; higher scores mean a worse outcome (higher scores indicate higher levels of sexual anxiety).

CONTACTS AND LOCATIONS:
Locations (1):
- Rey Juan Carlos University, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No